CLINICAL TRIAL: NCT06182423
Title: Chronic Pain Self-management for Older Adults With Cognitive Impairment: A Randomized Pilot Trial
Acronym: STEPS-CI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Mary Janevic, Research Associate Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00237064; R01AG071511-02S1 (NIH)
Record Dates: First submitted 2023-12-13; First posted 2023-12-26 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Chronic Pain; Cognitive Impairment
MeSH Terms: conditions — Chronic Pain; Cognitive Dysfunction | interventions — Palliative Care; Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- STEPS-CI Intervention Group (Experimental): Participants will engage in a behavioral intervention for chronic pain self-management that includes watching brief educational videos on a website and weekly sessions with a community health worker.
  Interventions: Behavioral: STEPS-CI (Support, Training, and Education for Pain Self-management- Cognitively Inclusive version)
- STEPS-CI Control Group (No Intervention): Members of the control group will not receive the STEPS-CI intervention. After completing the 8-week follow-up telephone survey, control group members will be invited to take part in a virtual workshop covering key STEPS-CI content and will receive program materials.

INTERVENTIONS:
Behavioral: STEPS-CI (Support, Training, and Education for Pain Self-management- Cognitively Inclusive version) — This intervention is a community health worker (CHW)-led chronic pain self-management program designed for older adults with chronic pain and mild to moderate cognitive impairment. It is a 7-week intervention that includes two primary components: a website that includes brief instructional videos on pain management skills as well as testimonials from individuals living with the two target health conditions; and weekly telephone sessions with a CHW to support and motivate participants in setting goals related to pain management. Reminder strategies and content addressing pain management challenges related to cognitive impairment are incorporated throughout. Participants may choose to work with a care partner during intervention activities.
  Arms: STEPS-CI Intervention Group

SUMMARY:
The goal of this randomized pilot trial is to test a chronic pain self-management program customized for people living with both chronic pain and cognitive impairment. The main questions it aims to answer are whether this program is feasible and acceptable, and whether it shows potential for improving pain-related outcomes. Intervention group participants will receive education and support from a community health worker in 7 weekly telephone sessions, and will watch a series of educational videos discussing a variety of chronic pain self-management skills. A control group will not receive the program, but after the final data collection point will be invited to attend a one-time remote session that summarizes intervention content, and will receive all program materials. Researchers will compare intervention and control groups after the program ends to see if the intervention group has less pain interference with daily activities.

ELIGIBILITY:
Inclusion Criteria:

* Age > 50 years;
* Have a cell or landline phone and internet access;
* Self-reported chronic musculoskeletal pain (pain in muscles or joints for > 3 months); >1 day/previous 30 when pain made it difficult to do usual activities.
* Self-reported mild cognitive impairment (MCI)/memory difficulties that at least sometimes interfere with usual daily activities

  * Willingness to meet by phone or video with a community health worker to learn potentially new ways to manage pain and commit to the duration of the program
  * Able to converse comfortably in English.

Exclusion Criteria:

* Serious acute illness or hospitalization in last month; planned major surgery in next three months that would interfere with program participation (e.g., knee replacement)
* Other issues that are judged by study team to preclude meaningful participation in study procedures (e.g. severe physical, cognitive, or psychiatric disorder).
* Current or prior participation in the parent STEPS study or the RESET (Re-Engaging in Self-Care and Enjoying Today) Study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2024-06-25 (Actual); Primary Completion 2025-06-11 (Actual); Study Completion 2025-06-11 (Actual)

PRIMARY OUTCOMES:
Change in pain interference | Baseline, 10 weeks from baseline
  The Pain Interference 6-item subscale of the Patient-Reported Outcomes Measurement Information System (PROMIS)-43 Adult Profile. Items ask how much pain in the last 7 days has interfered with daily activities such as household chores and social activities (1=not at all to 5=very much); raw total scale scores range from 6 (low interference) to 30 (high interference). When converted to T-scores (normed such that a score of 50 is the population mean and 10 T-score points=1 standard deviation), the possible range is 42 to 76, with a higher score representing a worse outcome.

SECONDARY OUTCOMES:
Change in pain intensity | Baseline, 10 weeks from baseline
  A numeric rating scale of pain in the last week ranging from 0 (no pain at all; best outcome) to 10 (worst pain you can imagine; worst outcome).
Change in subjective cognitive functioning | Baseline, 10 weeks from baseline
  The 4-item PROMIS Cognitive Function-Abilities Short Form 4a V. 2.0 measures perceived cognitive functioning in the last 4 days (e.g., "My mind has been as sharp as usual") on a scale from 1=not at all to 5=very much. Scores are converted to a standardized T-score metric, with a mean of 50 and a standard deviation of 10 in a referent population. A higher score means better cognitive functioning.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

DOCUMENTS (1):
  • Informed Consent Form (2024-05-20): https://cdn.clinicaltrials.gov/large-docs/23/NCT06182423/ICF_000.pdf